CLINICAL TRIAL: NCT03264950
Title: The Utility of Point Shear-wave Elastography to Assess for Hepatic & Pancreatic Fibrosis in Pediatric Cystic Fibrosis Patients
Brief Title: Utility of Point Shear-wave Elastography to Assess for Hepatic & Pancreatic Fibrosis in Pediatric CF Patients
Acronym: CFALD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Quais Mujawar, Pediatric Gastroenterologist, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B2017:077
Record Dates: First submitted 2017-06-23; First posted 2017-08-29 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-06

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis Liver Disease; Pancreatic Insufficiency Due to Cystic Fibrosis of Pancreas
MeSH Terms: conditions — Cystic Fibrosis | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Intervention Model Description: Patients (<18 years) will be recruited from from the Children's Hospital Winnipeg CF clinic. Charts will be reviewed for demographic and clinical data including blood work. Each patient will undergo shear wave elastography by a trained operator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIngle Arm (Other): All patients undergo Elastography. This is a single arm study
  Interventions: Diagnostic Test: Elastography

INTERVENTIONS:
Diagnostic Test: Elastography — an ultrasound exam after selecting the best acoustic window, a region of interest (ROI) is placed in an area of the liver perpendicular to the liver capsule, taking care not to include large vasculature or biliary structures.
  Similarly an acoustic window will be selected for the pancreas as well

SUMMARY:
Diagnosis of hepatic fibrosis is challenging as specific tests for detection of fibrosis in pediatric Cystic Fibrosis associated liver disease (CFALD) have not been developed and existing investigations do not correlate well with presence or severity of disease. Using a Liver biopsy it is difficult to diagnose this condition because of the patchy nature of the disease. Investigators intend to identify hepatic and pancreatic fibrosis in Cystic Fibrosis patients using Elastography and correlate this with their biochemical markers as well as histological findings of patients who have undergone liver biopsy for diagnosis of CFALD.

DETAILED DESCRIPTION:
Liver disease is increasingly common in cystic fibrosis (CF). As new therapeutic options emerge, life expectancy increases and common hepatobiliary manifestations impact on quality of life and survival of CF patients. Hepatobiliary abnormalities in CF vary in nature and range from defects attributable to the underlying CFTR gene defect to those related to systemic disease and malnutrition. Today complications of liver disease represent the third most frequent cause of disease-related death in patients with CF.

Cystic fibrosis-associated liver disease (CFALD) belongs to the group of common symptoms of this disease; however, due to the lack of specific and sensitive CFALD diagnostic markers, the epidemiological data may be incomplete. According to various sources, the prevalence rate of CFALD, diagnosed on the basis of clinical, biochemical and imaging (ultrasonography) tests, is 2-37% in children and young adults.

Cirrhosis is a final, irreversible stage of liver damage that leads to the failure of the organ. While liver biopsy is considered the gold standard to assess for Hepatic Fibrosis; it is invasive and potentially life threatening. The prognosis and management of chronic liver disease depends on the extent and progression of liver fibrosis, which constitutes the most important predictor of disease outcome.

The gold standard for diagnosis and staging of liver fibrosis has been liver biopsy. In addition to being an invasive procedure with potential complications of bleeding and severe pain, sampling error is an intrinsic problem due to the small sample size in a heterogeneous process.7,8 Inter-observer variability also limits diagnostic consistency.9-11 The development of several blood markers such as platelets, hyaluronic acid, type IV collagen, aminotransferase/platelet ratio index (APRI) and algorithm based serum models (Fibro Index, FIB-4, and Fibro Test) have been used but are affected by factors unrelated to the liver.

In the last decade, methods to noninvasively quantify liver fibrosis have been developed. The first available method was transient elastography (TE).It is a single-element ultrasound transducer operating at 5 MHz built on the axis of a piston like vibrator. By pushing a button, low-frequency (50 Hz) transient vibrations are transmitted, and the generated elastic shear waves propagate through underlying tissues. Pulse-echo ultrasound acquisitions are used to follow the propagation of the shear wave and to measure its velocity .

Several studies have demonstrated a high accuracy of TE in identifying significant fibrosis (F> 2) and cirrhosis (F= 4) in patients. It is a novel diagnostic tool that offers a rapid, non-invasive method for monitoring HF. The device measures liver stiffness by transmitting a vibration to determine the velocity of an elastic shear wave propagated through liver tissue.

Studies have documented utility of transient elastography in cystic fibrosis patients to assess hepatic fibrosis and secondary complications.

Newer modalities like Shear wave elastography techniques have been implemented in conventional real-time ultrasound systems, and several studies have shown their accuracy in the assessment of liver fibrosis. Shear wave elastography relies on the generation of shear waves determined by the displacement of tissues induced by the force of a focused ultrasound beam or by external pressure. The shear waves are lateral waves, with a motion perpendicular to the direction of the force that has generated them. They travel slowly (between 1 and 10 m/s) and are rapidly attenuated by tissue. The propagation velocity of the shear waves correlates with the elasticity of tissue .

Compared with TE, these techniques have the advantage of B-mode image guidance; thus, they can allow the user to choose the best acoustic window for correctly performing an examination in real time.

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years
* Confirmed diagnosis of cystic fibrosis attending Pediatric cystic fibrosis (CF) Clinic at Children's Hospital, Winnipeg.

Exclusion Criteria:

* Children with age >18 years

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-01-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the diagnostic properties of Shear wave Elastography | 6 months
  To evaluate the diagnostic properties of Shear wave Elastography (ElastPQ) in children with CF for detection of liver fibrosis.
  Investigators will look at the values of shearwave elastography and see how it correlates with the fibrosis values obtained on liver biopsy as well as with AST/platelet ratio index

SECONDARY OUTCOMES:
To compare findings/fibrosis of Transient Elastography vs ElastPQ | 6 months
  Investigators will compare degree of fibrosis on Transient Elastography vs Elast PQ to determine correlation .Some patients who have undergone liver biopsy will be correlated to liver fibrosis seen on biopsy.
  This will allow investigators to determine if Shear wave elastography can reliably detect fibrosis in patients with CFALD
To compare the pancreatic insufficiency/ fecal elastase and transient elastography from pancreas. | 6 months
  Investigators will see how well pancreatic fibrosis correlates with Fecal Elastase values and pancreatic endocrine function .
  This will let investigators know if Pancreatic elastography can help them in deciding which patients can have pancreatic insufficiency .

CONTACTS AND LOCATIONS:
Overall Officials: Quais Mujawar, Principal Investigator — University of Manitoba
Locations (1):
- Winnipeg Children's Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No